CLINICAL TRIAL: NCT00732563
Title: Radioguided Detection of Lymph Node Metastasis in Non-Small Cell Lung Cancer
Brief Title: Fludeoxyglucose F 18 in Detecting Lymph Node Metastasis in Patients With Stage I or Stage II Non-Small Cell Lung Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000601525; RPCI-I-97306
Record Dates: First submitted 2008-08-09; First posted 2008-08-12 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Lymph Node Excision; Neoadjuvant Therapy; Thoracic Surgical Procedures; Fluorodeoxyglucose F18; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: chemotherapy — Given IV and Orally
Procedure: lymphadenectomy — Removal of lymph nodes
Procedure: neoadjuvant therapy — Tumor reduction
Procedure: quality-of-life assessment — Correlative Study
Procedure: therapeutic conventional surgery — Treatment for cancer
Procedure: thoracic surgical procedure — removal of tissue
Radiation: fludeoxyglucose F 18 — given IV
Radiation: radiation therapy — undergoing radiotherapy

SUMMARY:
RATIONALE: Diagnostic procedures using fludeoxyglucose F 18 and a surgical probe may help find lymph node metastases in patients with early-stage non-small cell lung cancer.

PURPOSE: This clinical trial is studying how well fludeoxyglucose F 18 works in detecting lymph node metastasis in patients with stage I or stage II non-small cell lung cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the positive threshold of lymph node radioactivity after fludeoxyglucose F 18, utilizing the gamma probe, in patients with resectable stage I or II non-small cell lung cancer.
* Compare the accuracy of detecting thoracic lymph node metastases using positron emission tomography-computed tomography (PET-CT) versus the intra-operative hand-held gamma probe in these patients.
* Determine the ability of the gamma probe to detect lymph node micrometastases, resulting in upstaging in these patients.
* Assess the clinical relevance of the gamma probe-detected lymph node metastases by measuring patient survival, tumor recurrence, impact on patient quality of life, and cost.

OUTLINE: Patients undergo a positron emission tomography-computed tomography (PET-CT) scan within 90 days before surgery. Beginning 1-4 hours before surgery on day 1, patients receive an injection of fludeoxyglucose F 18 (FDG) and a mediastinoscopy is performed. FDG-avid lymph nodes are obtained and may undergo immunohistochemical analysis or standard analysis. Patients with mediastinal lymph node micrometastasis do not undergo primary tumor resection. Patients with ipsilateral mediastinal micrometastases undergo neoadjuvant chemotherapy prior to surgical resection. Patients with contralateral mediastinal micrometastases undergo definitive chemoradiotherapy. In the absence of mediastinal lymph node metastases (micro or macro), complete surgical resection is performed after the mediastinoscopy, including complete thoracic lymphadenectomy. The tumor and lymph nodes (both from mediastinoscopy and thoracotomy) undergo radioactivity measurements with the hand-held gamma probe. Fresh tumor and lymph node samples are stored for future studies.

Patients complete the Short Form 36 Health Survey (SF-36) before surgery and at 1, 3, and 6 months after surgery to assess the potential impact of the gamma probe on patient quality of life.

After completion of study, patients are followed every 6 months for 2 years, and then annually for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer

  * Stage I-II disease
  * Resectable disease
* Planning to undergo surgical resection
* No tumors that are not fludeoxyglucose F 18 (FDG)-avid on PET scan

PATIENT CHARACTERISTICS:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No previous allergic reaction to fludeoxyglucose F 18
* No contraindication to a pulmonary lobectomy and lymphadenectomy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-07-16 (Actual); Primary Completion 2012-06-29 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Survival rate at 2 years | 2 years
Recurrence rate at 2 years | 2 years

SECONDARY OUTCOMES:
Positive threshold of lymph node radioactivity | within 90 days
Comparison of the accuracy of detecting thoracic lymph node metastases using PET-CT scans versus intra-operative hand-held gamma probe | Within 90 days
Ability of the gamma probe to detect lymph node micrometastases, resulting in upstaging | Within 90 days
Quality of life | At 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chukwumere E. Nwogu, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States